CLINICAL TRIAL: NCT04687670
Title: Randomized Controlled Trial Comparing Personalized Embryo Transfer (pET) by the ERA Test Versus Conventional Frozen Embryo Transfer (FET) of Blastocysts in Infertile Women at Their First IVF/ICSI Cycle
Brief Title: RCT to Assess the Clinical Benefit of the ERA Test in Infertile Women at Their First IVF/ICSI Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: RenJi Hospital (Other); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PUTH ERA 1.0
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-04

CONDITIONS: Infertility, Female; IVF/ICSI
Keywords: Personalized Embryo Transfer; Endometrial Receptivity Analysis; Conventional Frozen Embryo Transfer; Randomized Controlled Trial
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group(pET) (Experimental): Personalized embryo transfer of a single vitrified blastocyst in a HRT cycle according to the ERA test results.
  Interventions: Diagnostic Test: ERA
- Control group(FET) (Active Comparator): Frozen embryo transfer of a single vitrified blastocyst in a HRT cycle according to the clinical standard practice.
  Interventions: Diagnostic Test: ERA

INTERVENTIONS:
Diagnostic Test: ERA — Before the randomization, Endometrial Fluid (EF) and Endometrial Biopsy (EB) samples will be collected from all participants. EF will be obtained by aspiration immediately prior to the EB after around 120 hours of progesterone (P) impregnation following the standard HRT cycle. The results of the ERA test will be provided to participants and their gynecologists for the personalized embryo transfer.
  Arms: Intervention group(pET)
Diagnostic Test: ERA — Before the randomization, Endometrial Fluid (EF) and Endometrial Biopsy (EB) samples will be collected from all participants. EF will be obtained by aspiration immediately prior to the EB after around 120 hours of progesterone (P) impregnation following the standard HRT cycle. The results of the diagnosis will not be disclosed with the patients randomized into this arm nor with their gynecologists.
  Arms: Control group(FET)

SUMMARY:
Endometrial receptivity takes place in a self-limited period of time during the endometrial mid-secretory stage. This period, named as window of implantation (WOI), is modulated by molecular changes allowing embryo implantation to take place.

It has been already demonstrated the existence of transcriptomic profiles that are characteristics of each endometrial phase: pre-receptive, receptive and post-receptive. 'Igenomix' group developed a molecular tool able to classify the endometrium based on its transcriptomic profile, the Endometrial Receptivity Analysis (ERA). This molecular tool analyses, by next generation sequencing (NGS), the expression of 248 genes related to implantation coupled to a computational predictor to identify the specific transcriptomic profile for each endometrial stage. This test has been applied at clinical level from 2010, helping to synchronize a viable embryo with a receptive endometrium through the personalized embryo transfer (pET). It aims to improve clinical implantation by personalizing, diagnosing, and synchronizing the endometrial factor.

Our goal in this project is to investigate at what extent, if any, the analysis of the endometrial factor, at receptivity level, in patients at their first in vitro fertilization (IVF) cycle improves their clinical outcome through a personalized embryo transfer by the ERA test in comparison to embryo transfer(FET).

DETAILED DESCRIPTION:
When the transcriptomic signature of human endometrial receptivity was reported, Igenomix developed the ERA, a molecular tool able to diagnose the endometrial receptivity by NGS and a computational predictor. The accuracy of this diagnostic tool has been shown to be superior to endometrial histology, and its results are reproducible 29 to 40 months later.

The ERA test allows to transfer in a personalized manner by synchronizing the embryo with the WOI of the patient. Nowadays, it has been published that around 30% of patients present 1 or 2 days of displacements and about 50% show 12 hours of displacement.

The ERA has been broadly applied around the world in order to increase the probabilities of recurrent implantation failure patients becoming pregnant. Recently, a multicenter international open-label randomized controlled trial comparing personalized embryo transfer guided by the ERA test versus frozen and fresh embryo transfer was carried out at first appointment of infertile patients undergoing IVF. The current project aims to assess in a randomized way the potential improvement on the clinical outcome of Chinese infertile patients at their first IVF cycle by diagnosing, personalizing and synchronizing the endometrial factor with the ERA. To do that, only the outcomes of the first single embryo transfers performed after the inclusion of each patient will be considered.

Considering a 30% of possible drop-outs, a total of 714 patients will be recruited (357 randomized in each group). They will be allocated on a balanced way (assigned by chance like the flip of a coin) in one of the two arms described below. Reproductive outcomes (defined following The International Glossary on Infertility and Fertility Care, 2017) will be compared between the two groups.

Data exported from the source documents will be duly codified and treated in order to protect the clinical and personal information of participants in accordance with the current local legislation.

All the statistical analysis performed on the data, as well as the procedures, will be registered in a detailed Statistical Analysis Plan (SAP) that will be developed during the study and before starting data analysis.

An interim analysis of this data is planned once 50% of the recruitment has been achieved. Besides and at that same moment, the study will be overseen by an independent Data Monitoring Committee.

All the statistical procedures will be done systematically by both, intention to treat analysis (ITT) and per protocol analysis (PP). The ITT analysis will include all randomized patients recruited and assigned to one of two groups after endometrial biopsy collection. The PP analysis will be applied to those patients who adequately follow the protocol assigned according to their group and arm and in whom the transfer of the good quality blastocyst is performed.

ELIGIBILITY:
Inclusion criteria:

* Patients whose written ICF approved by the EC has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
* Patients undergoing their first IVF/ICSI cycle (first oocyte pick up, freezing all) with their own oocytes that will receive single embryo transfer of frozen blastocyst stage embryos (day 5/6) on an HRT cycle.
* At least 2 morphologically good quality embryos already vitrified in blastocyst stage (day 5/6).
* Maternal Age: ≤37 years to rule out embryo factor in aging patients.
* BMI: 18.5 - 30.0 kg / m2 (both inclusive).
* Normal ovarian reserve (defined as: AFC ≥ 8; AMH level ≥1.0 ng/ml and/or FSH < 8 mU/ml) before the controlled ovarian stimulation (COS) initiation.
* Serum P levels ≤ 1.5 ng/ml, measured within 24 hours before the hCG administration in the COS cycle.
* Negative serological tests for HIV, HBV, HCV, RPR.

Exclusion criteria:

* Patients with repeated miscarriages (> 2 previous biochemical pregnancies or > 2 spontaneous miscarriages).
* Male partner with severe male factor (spermatozoa < 2 million/ml). Semen donor is allowed.
* Patients who are intrauterine device (IUD) carriers in the last 3 months before sample collection.
* Adenomyosis or any pathological finding affecting the endometrial cavity such as polyps/sub-mucosal myomas, intramural myomas > 4 cm, or hydrosalpinx must be previously operated at least 3 months before the endometrial samples are obtained. (Note: Patients are allowed to participate if the pathology is corrected before performing any study procedure).
* Embryos analysed using preimplantation genetic testing for aneuploidies (PGT-A).
* Any illness or medical condition that is unstable or affect the safety of the patient and compliance of the study.

Max Age: 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 714 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | From date of embryo transfer until 40 weeks
  The number of deliveries that resulted in at least one live birth per ET (transferred patient). Live birth is defined as the complete expulsion or extraction from a woman of a product of conception after 22 weeks of gestation, which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached.

SECONDARY OUTCOMES:
Implantation rate | From date of embryo transfer until 5-6 weeks
  The number of gestational sacs observed by vaginal ultrasound at the 5th gestational week divided by the number of embryos transferred.
Clinical miscarriage rate | From date of embryo transfer until 20 weeks
  Number of spontaneous pregnancy losses in which a gestational sac/s was previously observed, per number of pregnancies.
Biochemical pregnancy rate | From date of embryo transfer until 5-6 weeks
  Number of pregnancies diagnosed only by βhCG detection without a gestational sac visualized by vaginal ultrasound at the 5th week of pregnancy, per number of pregnancies.
Ectopic pregnancy rate | From date of embryo transfer until 8 weeks
  Number of pregnancies outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology, per number of pregnancies.
Incidence of WOI displacement in the study population | From date of randomization until 1-2 months
  Number of patients with the WOI displaced during their participation
pregnancy rate | From date of embryo transfer until 2 weeks
  Pregnancy rate is the number of patients with positive serum level of beta-HCG per embryo transfer.
Obstetric complications | From date of embryo transfer until 40 weeks
  Type and number of obstetric complications during pregnancy
Delivery complications | From date of embryo transfer until 40 weeks
  Type and number of delivery complications
Cost-effectiveness between pET and FET groups | 2 years
  To estimate the average cost per patient in each treatment to achieve a live newborn.

OTHER OUTCOMES:
ERA test validation in endometrial fluid | From date of randomization until 1-2 months
  Clinical validation of a non-invasive endometrial receptivity test diagnosis by comparing results from endometrial biopsy and fluid

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Principal Investigator — Peking University Third Hospital, Beijing
Locations (3):
- China (3):
  - Northwest Women's and Children's Hospital, Xi'an, Shaanxi
  - Peking University Third Hospital, Beijing
  - Renji Hospital, Shanghai